CLINICAL TRIAL: NCT02091791
Title: High Versus Low Level of Lumbar Traction in Acute Lumbar Sciatica Due to Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2754
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Lumbar Sciatica Secondary to Disc Herniation
Keywords: acute lumbar sciatica, lumbar traction, traction force, radicular pain, lumbar functional parameters, disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LT10 (Experimental): Long duration (30 minutes) traction sessions of "low force" (10% of body weight) for 2 weeks (5 sessions/week).
  Interventions: Procedure: Traction sessions
- LT50 (Experimental): Long duration (30 minutes) traction sessions of "high force" (50% of body weight) for 2 weeks (5 sessions/week).
  Interventions: Procedure: Traction sessions

INTERVENTIONS:
Procedure: Traction sessions
  Other Names: Traction sessions using a spinal traction system

SUMMARY:
The aim of this study is to compare two levels (high and low forces) of short term lumbar traction on pain and functional tests of the lower limbs in a specific population of patients presenting with acute lumbar sciatica secondary to disc herniation. The investigators hypothesize that, in this particular medical condition, high level of lumbar traction might be more effective than low level lumbar traction in decreasing the pain associated with acute sciatica.

ELIGIBILITY:
Inclusion Criteria:

* less than 6-week lumbar sciatica secondary to disc herniation, confirmed by pain radiating down the leg along the distribution of the sciatic nerve together with positive straight leg raising test (SLRT)

Exclusion Criteria:

* symptoms persisting for more than 6 weeks
* signs of clinical neurological deficit
* lumbar sciatica not caused by disc herniation
* presence of lumbar tomodensitometry abnormalities
* Subjects younger than 18
* pregnant women
* patients on medical leave for more than 3 weeks at inclusion
* patients with history of lumbar surgery
* patients who already had lumbar traction therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in radicular pain graduated from 0 to 100 mm | Measurement of radicular pain using a visual analogue scale (VAS) At baseline (day 0 - D0) as well as at day 14 (D14) (end of treatment) and day 28 (D28) (after 2 weeks follow-up).

SECONDARY OUTCOMES:
Global mobility of the lumbar-pelvic spine evaluated using the finger to toe test (FTT, in cm) | At baseline (day 0 - D0) as well as at day 14 (D14) (end of treatment) and day 28 (D28) (after 2 weeks follow-up).
Lumbar spine mobility (in mm) assessed with the Schöber-Macrae's test | At baseline (day 0 - D0) as well as at day 14 (D14) (end of treatment) and day 28 (D28) (after 2 weeks follow-up).
Signs of nerve root compression evaluation assessed by the SLRT and EIFEL score | At baseline (day 0 - D0) as well as at day 14 (D14) (end of treatment) and day 28 (D28) (after 2 weeks follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Eve ISNER-HOROBETI, MD, Principal Investigator — Institut Universitaire de Réadaptation Clémenceau - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Médecine Physique et de Réadaptation, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg, France

REFERENCES:
- [Result] Isner-Horobeti ME, Dufour SP, Schaeffer M, Sauleau E, Vautravers P, Lecocq J, Dupeyron A. High-Force Versus Low-Force Lumbar Traction in Acute Lumbar Sciatica Due to Disc Herniation: A Preliminary Randomized Trial. J Manipulative Physiol Ther. 2016 Nov-Dec;39(9):645-654. doi: 10.1016/j.jmpt.2016.09.006. Epub 2016 Nov 9. PMID 27838140